CLINICAL TRIAL: NCT05063435
Title: Cardiovascular Structure and Function in the Mucopolysaccharidoses
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital of Orange County (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 200107
Record Dates: First submitted 2021-07-15; First posted 2021-10-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Mucopolysaccharidoses; Carotid Disease; Cardiac Disease; Inflammation
Keywords: mucopolysaccharidosis; carotid; cardiac; cardiovascular; biomarker; longitudinal; observational
MeSH Terms: conditions — Mucopolysaccharidoses; Heart Diseases; Inflammation | interventions — Ultrasonography, Carotid Arteries; Echocardiography; Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Carotid ultrasonography — 1. Study takes 10 - 15 minutes to complete
  2. Subject will be asked to lay still and quietly during procedure
  3. The ultrasound probe will be placed on one side of the neck to capture images of the carotid artery. When images from one side have been captured, the probe will be moved to the other side of the neck to capture images from the other carotid artery.
  4. Blood pressure and heart rate will be obtained during the study
  5. Results will be anonymized, digitized and stored on CD with unique identifier
  Other Names: Carotid ultrasound
Diagnostic Test: Echocardiography, transthoracic — 1. Study takes 15 - 20 minutes to complete
  2. Subject will be asked to lay still and quietly during procedure
  3. The technician will apply an ultrasound probe to the chest. Images and movies will be acquired.
  4. Results will be digitized and stored on CD
  Other Names: Echocardiogram
Procedure: Venipuncture — 1. 10 mL of blood total will be drawn (5 mL in a blue top citrate tube, 5 mL in a purple top EDTA tube). Measurements of cytokines, clusterin, lipidomics, cathepsin S protease, and elastin (previously identified potential biomarker candidates) will be performed.
  2. Blood will preferably be drawn via venipuncture, but if patient has a port-a-cath already implanted and is having blood drawn via port-a-cath for clinically required reasons, then study-related blood draw via port-a-cath can take place concurrently with clinically required blood draws.
  Other Names: Blood draw; Phlebotomy

SUMMARY:
This study's investigators previously demonstrated the potential utility of non-invasive carotid ultrasonography to calculate carotid intima media thickness (cIMT) and stiffness (as measured by the three parameters, carotid cross-sectional distensibility [cCSD], carotid cross-sectional compliance [cCSC], and carotid incremental elastic modulus [cIEM]) in people with mucopolysaccharidoses (MPS).

Investigators also studied arterial gene expression in animal models of MPS, and identified upregulation of a number of markers potentially tied to atherosclerosis and inflammation. These include the atherosclerotic marker known as Clusterin (CLU), Cathepsin S, Elastin, and the inflammatory cytokines interleukin 1-α, interleukin 1-β, interleukin 2, and interleukin 6. Other studies have identified elevation in circulating tumor necrosis factor-α correlating with pain and physical disability in certain mucopolysaccharidoses.

Since these studies are cross sectional, and not longitudinal, this study aims to annually measure these previously studied biomarkers (carotid measurements, circulating cytokines, cathepsin S, elastin, and CLU) in a large cohort of MPS patients. This study is a 3-year, prospective, anonymized, longitudinal assessment of cardiovascular structure, function, and circulating biomarkers in patients with mucopolysaccharidoses.

DETAILED DESCRIPTION:
Specific Aims

1. Annually assess cardiac and carotid structure and function utilizing ultrasonography, in patients with mucopolysaccharidoses
2. Annually measure circulating levels of clusterin, elastin, cathepsin S, lipids, and cytokines in patients with mucopolysaccharidoses

Target enrollment 30 subjects at CHOC Children's Hospital

Study Protocol

Screening

1. Study Investigators will identify eligible patients to participate in the study from their current patient population and future referrals.
2. Eligible patients will be provided with study information on the study during their standard of care metabolic clinic visit.

Informed Consent

1. Informed consent will be obtained following the requirements set forth by 21 CFR 50.25.
2. Patients interested in the study will be provided the informed consent document. The document will be reviewed in a private quiet room and ample time for questions will be provided. The patient can keep a copy of the consent if they wish to discuss the study with friends and family. Consent will only be obtained once the patient has had time to ask questions and is aware that the study is completely voluntary.

Initial entry

1. Information regarding age, sex, MPS diagnosis (including genetic mutation and enzymatic levels, if possible) will be obtained
2. Height and weight will be obtained. If patient has had a recent (within 3 months) evaluation at CHOC Children's with height and weight, those parameters may be used
3. Medical records will be obtained specifically focusing upon

   1. the genetic and/or enzymatic testing used to confirm the MPS diagnosis
   2. the treatment status (treated or not) and duration of treatment (calculated by the difference between date of first carotid imaging and date of first treatment)
4. Carotid ultrasonography will be obtained

   1. Study takes 10 - 15 minutes to complete
   2. Subject will be asked to lay still and quietly during procedure
   3. Blood pressure and heart rate will be obtained during the study
   4. Results will be digitized and stored on CD
5. Echocardiography will be obtained

   1. Study takes 15 - 20 minutes to complete
   2. Subject will be asked to lay still and quietly during procedure
   3. Results will be digitized and stored on CD
6. Venipuncture / phlebotomy

   1. 10 mL of blood total will be drawn (5 mL in a blue top citrate tube, 5 mL in a purple top EDTA tube). Measurements of cytokines, clusterin, lipidomics, cathepsin S protease, and elastin (previously identified potential biomarker candidates) will be performed.
   2. Blood will preferably be drawn via venipuncture, but if patient has a port-a-cath already implanted and is having blood drawn via port-a-cath for clinically required reasons, then study-related blood draw via port-a-cath can take place concurrently with clinically required blood draws.

Annual studies Procedures 2), 4), 5), and 6) will be repeated on an annual basis for a total of three years

ELIGIBILITY:
Inclusion Criteria:

1. Any patient with a molecularly confirmed diagnosis of mucopolysaccharidosis is eligible to enroll in this study
2. Parental / patient informed consent

Exclusion Criteria:

1. Any reason that the investigators would deem a patient unable to participate in this study
2. Inability to participate in the assessments required for this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with a diagnosis of mucopolysaccharidosis who provides informed consent is eligible for this study. Mucopolysaccharidoses are a group of inherited metabolic disorders involving abnormal degradation of glycosaminoglycans. There are 11 different genes which, when altered, can give rise to a mucopolysaccharidosis. People with this diagnosis can develop significant cardiovascular disease (left ventricular hypertrophy, valvular dysfunction, aortic root dilatation, arterial wall thickening and stiffness).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-10-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Event | 3 years
  A cardiovascular event is defined by new onset of clinically significant aortic or mitral valve disease, aortic root dilatation, cardiomyopathy, reduction in cardiac contractile function, myocardial ischemia, myocardial infarction, or cerebrovascular accident

SECONDARY OUTCOMES:
Age | 3 years
  Change of age of subject (unit: years)
Height | 3 years
  Change of height of subject (unit: meters)
Weight | 3 years
  Change of weight of subject (unit: kilograms)
Blood pressure | 3 years
  Change in systolic and diastolic blood pressure over the duration of the study (unit: millimeters of mercury)
Carotid structure | 3 years
  Change in carotid intima media thickness over the duration of the study (mm).
Carotid stiffness | 3 years
  Change in carotid cross-sectional distensibility over the duration of the study (unit: %). This metric is acquired in the carotid ultrasound, and measures the stiffness of the carotid artery via quantitation of the difference between end-systolic and end-diastolic carotid diameter.
Cardiac structure (left ventricle) | 3 years
  Change in left ventricular mass index over the duration of the study (unit: grams / m2 body surface area). This metric is acquired in the echocardiogram, and quantitates the amount of myocardium in the left ventricle.
Cardiac structure (aortic root diameter) | 3 years
  Change in aortic root measurement over the duration of the study (unit: mm). This metric is acquired in the echocardiogram, and quantitates the width of the aortic root.
Mitral valve function | 3 years
  Assessment of changes in mitral valve function over the duration of the study (unit: 4 point Likert scale from 0 [none] to 4 [severe]). This metric is acquired during the echocardiogram, and assess the degree of mitral valve insufficiency.
Aortic valve function | 3 years
  Assessment of changes in aortic valve function over the duration of the study (unit: 4 point Likert scale from 0 [none] to 4 [severe]). This metric is acquired during the echocardiogram, and assess the degree of aortic valve insufficiency.
Inflammatory biomarkers (Tumor Necrosis Factor - alpha) | 3 years
  Change in plasma TNFa over the duration of the study.
Inflammatory biomarkers (Cathepsin S) | 3 years
  Change in plasma Cathepsin S over the duration of the study. (Unit: mcg/L)
Inflammatory biomarkers (Elastin) | 3 years
  Change in plasma Elastin levels over the duration of the study. (Unit: ng/mL)
Inflammatory biomarkers (Clusterin) | 3 years
  Change in plasma clusterin levels over the duration of the study. (Unit: mcg/mL)
Inflammatory biomarkers (lipidomics) | 3 years
  Change in plasma lipid levels over the duration of the study. (Unit: mcmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Wang, M.D., Principal Investigator — CHOC Children's Hospital
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No
Since we are the sole site, we do not have any plans to share individual data at this point. Once the study has completed data collection and analysis, data will be shared in aggregate.

REFERENCES:
- [Background] Wang RY, Covault KK, Halcrow EM, Gardner AJ, Cao X, Newcomb RL, Dauben RD, Chang AC. Carotid intima-media thickness is increased in patients with mucopolysaccharidoses. Mol Genet Metab. 2011 Dec;104(4):592-6. doi: 10.1016/j.ymgme.2011.09.004. Epub 2011 Sep 10. PMID 21963080
- [Background] Wang RY, Braunlin EA, Rudser KD, Dengel DR, Metzig AM, Covault KK, Polgreen LE, Shapiro E, Steinberger J, Kelly AS. Carotid intima-media thickness is increased in patients with treated mucopolysaccharidosis types I and II, and correlates with arterial stiffness. Mol Genet Metab. 2014 Feb;111(2):128-32. doi: 10.1016/j.ymgme.2013.11.001. Epub 2013 Nov 12. PMID 24268528
- [Background] Wang RY, Rudser KD, Dengel DR, Braunlin EA, Steinberger J, Jacobs DR, Sinaiko AR, Kelly AS. The Carotid Intima-Media Thickness and Arterial Stiffness of Pediatric Mucopolysaccharidosis Patients Are Increased Compared to Both Pediatric and Adult Controls. Int J Mol Sci. 2017 Mar 15;18(3):637. doi: 10.3390/ijms18030637. PMID 28294991
- [Background] Wang RY, Rudser KD, Dengel DR, Evanoff N, Steinberger J, Movsesyan N, Garrett R, Christensen K, Boylan D, Braddock SR, Shinawi M, Gan Q, Montano AM. Abnormally increased carotid intima media-thickness and elasticity in patients with Morquio A disease. Orphanet J Rare Dis. 2020 Mar 17;15(1):73. doi: 10.1186/s13023-020-1331-y. PMID 32183856